# Evaluation of the analgesic efficacy of the combination of deksketoprofen + paracetamol and the combination of naproxen sodium + codeine in patients with acute dental pain

İbrahim Doğru<sup>1</sup>, Levent Ciğerim <sup>1</sup>

<sup>1</sup> Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial

Surgery, Van, TURKEY

Corresponding author: İbrahim Doğru

Address: Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial

Surgery, Van, Turkey Postal Code: 65080

E-mail address: <u>ibrahimdogru@yyu.edu.tr</u> Phone:+905418952655 Office Phone: 904322251744

Fax: +904322251747

#### İbrahim DOĞRU

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery <a href="mailto:ibrahimdogru@yyu.edu.tr">ibrahimdogru@yyu.edu.tr</a>, +905418952655, <a href="https://orcid.org/0000-0001-9174-9401">https://orcid.org/0000-0001-9174-9401</a>

### Levent CİĞERİM

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery leventcigerim@yyu.edu.tr, +905321633287, https://orcid.org/0000-0001-5218-8568

## Study Protocol, Methods and Procedures to be Applied:

The study is planned to be carried out on 90 patients aged 18 and over, who applied to Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, with complaints of acute pericoronitis caused by lower half impacted wisdom teeth. When patients first apply to the clinic, their anamnesis and demographic information will be obtained through anamnesis form. Patients who meet the inclusion criteria and volunteer will be included in the study.

Patients will be randomly divided into 2 groups. Medications will be given to patients by auxiliary staff and the study will be double-blind. Group A (active control group) received 550 mg naproxen sodium + 30 mg codeine phosphate and group B (research group) received 25 mg dexketoprofen trometamol + 300 mg paracetamol 2 times daily for 7 days; and amoxicillin 500 mg 3 times daily for 5 days in addition to analgesics for infection control due to acute pericoronitis. Paracetamol 500 mg was administered as rescue medication. Patients were instructed not to take rescue medication unless they had to and, if they did, to record the time and number of doses on the form given to them. Patients in the study groups received the first dose of the drugs from us and continued to receive subsequent doses every 12 hours.

A Visual Analogue Scale (VAS) with numbers ranging from 0 - no pain to 10 - unbearable pain was used to assess pain. Patients were asked to record their VAS score on the form at the 6th hour (T1), 12th hour (T2), 18th hour (T3), 24th hour (T4), 2nd day (T5), 3rd day (T6), 4th day (T7), 5th day (T8), 6th day (T9) and 7th day (T10) after the first dose (T0 of study drug.

Obtained data will be analyzed and evaluated statistically.

### **Statistical Data Analysis:**

Descriptive statistics for continuous variables in our study; As Average, Standard Deviation, Minimum and Maximum values; will be expressed as numbers and percentages for categorical variables. Mann-Whitney U analysis will be used to compare group means in terms of continuous independent variables. In addition, the Wicoxon test will be calculated in the comparison of double dependent groups. In order to determine the relationship between these variables, Spearman correlation coefficients will be calculated separately for the groups. Chi-square test will be used to determine the relationship between groups and categorical variables. Statistical significance level will be taken as 5% in calculations and SPSS statistical package program will be used for calculations.